CLINICAL TRIAL: NCT04253652
Title: Investigating the Effects of Iron on the Gastrointestinal Tract
Acronym: GI-iron
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Functional Gut Clinic (Other)
Collaborators: Anglia Ruskin University (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Consultant Clinical Scientist, The Functional Gut Clinic
Other Study IDs: FGC19002
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Iron Deficiency Anemia; Constipation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral iron: These patients will have diagnosed with iron deficiency anaemia and been prescribed oral iron supplements as part of their treatment from their doctor. This will be in accordance with the NICE guidelines; 200mg capsules containing 65mg elemental iron, 2-3 times a day for a period of atleast 1 month.
  Interventions: Other: Fasted breath samples; Other: IBS-SSS; Other: Daily diary; Other: Exploratory research: stool samples
- Intravenous iron: These patients will have diagnosed with iron deficiency anaemia and been prescribed intravenous iron as part of their treatment from their doctor. Participants will receive an infusion of either 1000mg or 1500mg
  Interventions: Other: Fasted breath samples; Other: IBS-SSS; Other: Daily diary; Other: Exploratory research: stool samples

INTERVENTIONS:
Other: Fasted breath samples — Will be completed pre and post iron therapy
Other: IBS-SSS — Will be completed pre and post iron therapy
Other: Daily diary — Monitoring stool form, consistency and frequency on a daily basis for 4 weeks
Other: Exploratory research: stool samples — Completed pre and post iron therapy for a subset of patients enrolled in the study

SUMMARY:
Many patients that are prescribed iron report gastrointestinal side effects. This research project aims to investigate if the gastrointestinal symptoms of taking iron supplementation are related to changes in gases produced by bacteria in the gastrointestinal tract.

DETAILED DESCRIPTION:
This study is a pre-post interventional, two armed prospective cohort study where patients who are newly diagnosed with iron deficiency anaemia are prescribed iron therapy (either oral iron supplements, 200mg capsules containing 65mg of iron 2-3 times daily, or intravenous iron 1000-1500mg) as part of their standard care. Participants will be asked to provide breath samples and complete the IBS-SSS questionnaire at baseline and after 4 weeks of taking the iron therapy as part of their standard care. A diary including stool consistency and frequency will also be completed by participants on a daily basis. For further exploratory research, some participants from each the oral and IV iron arm will be asked to provide stool samples at baseline and 4-weeks post iron therapy to assess any microbiome changes in response to iron therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Male or non-pregnant female and is age 18 years to 80 years.
3. Can communicate well with the Investigator and to comply with the requirements for the entire study.
4. Capacity to understand written English.
5. New diagnosis iron-deficient anaemia.
6. Prescribed IV iron therapy or oral iron supplementation which contains 65mg elemental iron, two or three times per day for a period of at least 1 month or, will receive 1000mg or 1500mg of intravenous iron, as part of their standard care.
7. Participant agrees to wait until after taking baseline breath samples and completing the IBS-SSS questionnaire before starting their iron therapy.
8. Participant agrees to follow pre-test diet for 24 hours before giving test sample.
9. Participant agrees to refrain from strenuous physical activity on the day of the breath test.
10. Refrain from smoking on the day of the breath test.
11. Agree to complete an overnight fast on the night before the breath test. Food and drink must be withheld until after all breath test samples have been taken.
12. No probiotics for 14 days before the breath test or during the study.
13. Body mass index between 18.5 and 34.9kg/m2 (bounds included).
14. Not antibiotics for 4-weeks before the start of the study or during the study

Exclusion Criteria:

1. Using an opioid based medication.
2. Antibiotics in the 4 weeks prior to enrolment.
3. Colonoscopy/sigmoidoscopy in the 1 week prior to enrolment, unless they have taken their baseline breath sample and IBS-SSS questionnaire before completing the required bowel preparation.
4. Diagnosis of any organic gastrointestinal disease, including inflammatory bowel disease, coeliac disease and diverticulitis.
5. Mechanical obstruction of the GI tract.
6. Participant is diabetic.
7. Participant has any hepatic disease.
8. Participant has any disease of the CNS.
9. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or sponsor member.
10. Previous abdominal or colorectal surgery except appendectomy, cholecystectomy, or hysterectomy.
11. Participant has had iron therapy in the 12 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 oral iron participants 55 IV iron participants
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2023-03-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Breath | 4 weeks apart
  Difference in methane levels in breath samples from baseline and 4-weeks since commencing iron therapy. This will be measured in parts per million (ppm).

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | 4 weeks apart
  Comparison in change of IBS-SSS score from baseline to 4 weeks since commencing iron therapy. The minimum score is 0 and maximum score is 500. The greater the score, the worse the severity and frequency of symptoms of abdominal pain and distention, and increased dissatisfaction of overall bowel functioning.
Stool consistency | 4 weeks apart
  Change in stool frequency and form according to the bristol stool chart and abdominal symptoms during the 4 weeks since commencing iron therapy.

OTHER OUTCOMES:
Exploratory | 4 weeks apart
  Qualitative and Quantitative data for faecal microorganisms at baseline and 4-weeks since commencing iron therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, Principal Investigator — The Functional Gut Clinic
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No